CLINICAL TRIAL: NCT07388485
Title: The Effect of an Interactive Digital Art-Based Relaxation Program on Physiological Parameters, Anxiety, and Emotional Distress in Children Receiving Treatment in the Pediatric Intensive Care Unit: A Randomized Controlled Trial
Brief Title: Interactive Digital Art-Based Relaxation Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Hazal Ozdemir Koyu, Dr. Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-2215
Record Dates: First submitted 2026-01-15; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Critical Illness; Anxiety
Keywords: Pediatric Intensive Care Unit; Children; Interactive Digital Art-Based Relaxation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a parallel-group randomized controlled trial. Eligible participants will be randomly assigned in a 1:1 ratio to either the intervention group or the control group. The intervention group will receive an interactive digital art-based relaxation program in addition to standard pediatric intensive care, while the control group will receive standard pediatric intensive care alone. Outcomes will be assessed at baseline and after completion of the intervention, with no crossover between groups.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants and intervention providers cannot be blinded. However, outcome assessment will be performed by a researcher who is blinded to group allocation. The outcome assessor will not be involved in the intervention delivery and will be unaware of participants' group assignments to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Received Standard Care
- Intervention Group (Experimental): Received Interactive Digital Art-Based Relaxation Program
  Interventions: Other: Interactive Digital Art-Based Relaxation Program

INTERVENTIONS:
Other: Interactive Digital Art-Based Relaxation Program — The Interactive Digital Art-Based Relaxation Program is a nurse-guided, technology-assisted psychosocial intervention designed for children aged 7-12 years receiving care in the pediatric intensive care unit. The program consists of three individual sessions delivered via a tablet device. Each session lasts approximately 8-10 minutes and integrates interactive digital art activities with guided breathing, emotional awareness, and relaxation techniques.
  During the sessions, children are encouraged to engage in simple digital art creation (e.g., drawing, color selection, and visual expression) while following age-appropriate breathing and relaxation prompts provided by the nurse. The intervention is designed to promote emotional expression, reduce anxiety, and support physiological stabilization by facilitating relaxation and emotional regulation. All sessions are conducted at the bedside under nurse supervision and are tailored to the child's clinical condition and tolerance.
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial aims to evaluate the effects of an Interactive Digital Art-Based Relaxation Program on physiological parameters, anxiety levels, and emotional distress in children aged 7-12 years receiving care in a pediatric intensive care unit (PICU). Children in the intervention group will receive three short, nurse-guided digital art-based relaxation sessions delivered via tablet, while the control group will receive standard PICU nursing care. Outcomes will be assessed using physiological measurements and validated psychological assessment tools before and after the intervention.

DETAILED DESCRIPTION:
Children hospitalized in pediatric intensive care units are exposed to multiple stressors, including invasive procedures, environmental noise, physical discomfort, and separation from family members. These factors may lead to increased anxiety, emotional distress, and physiological dysregulation, even in children who are conscious and not receiving sedation. There is a growing need for brief, feasible, and child-friendly non-pharmacological interventions that can be safely implemented in the PICU setting to support emotional well-being and physiological stability.

This study is designed as a parallel-group, randomized controlled trial to evaluate the effectiveness of an Interactive Digital Art-Based Relaxation Program in reducing anxiety and emotional distress and improving physiological parameters in children aged 7-12 years receiving care in a pediatric intensive care unit. The study will be conducted between February 2026 and March 2027 in the Pediatric Intensive Care Unit of Etlik City Hospital, Ministry of Health.

A total of 60 children who meet the inclusion criteria will be randomly assigned to either the intervention group (n = 30) or the control group (n = 30) using simple randomization. Randomization will be performed by an independent statistician using a computerized randomization tool. Eligible participants will be conscious, hemodynamically stable, not receiving continuous sedative or analgesic infusion, and able to follow verbal instructions.

Children in the intervention group will receive an Interactive Digital Art-Based Relaxation Program consisting of three sessions. Each session will last approximately 8-10 minutes and will be delivered via a tablet under nurse guidance. The program integrates interactive digital art activities with relaxation components designed to promote emotional expression, attention regulation, and calming responses. The control group will receive standard pediatric intensive care nursing care without additional psychosocial intervention.

Data will be collected at baseline and after completion of the intervention. Baseline assessments will include a descriptive characteristics form, physiological parameters (heart rate, respiratory rate, blood pressure, oxygen saturation, and pain), the State Anxiety Inventory for Children, and the Emotion Thermometer. Physiological parameters will also be recorded immediately before and after each intervention session. Post-intervention assessments will include repeated physiological measurements, the State Anxiety Inventory for Children, and the Emotion Thermometer.

The primary outcomes of the study are changes in physiological parameters and anxiety levels. Secondary outcomes include changes in emotional distress levels. It is hypothesized that children who participate in the Interactive Digital Art-Based Relaxation Program will demonstrate improved physiological stability, reduced anxiety, and lower emotional distress compared to those receiving standard care.

The findings of this study are expected to contribute to evidence-based pediatric intensive care nursing practices by providing support for the integration of short, technology-assisted, art-based psychosocial interventions into routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* • Be between 7 and 12 years of age

  * Be conscious and able to respond to commands
  * Not be receiving sedative/analgesic infusion or be at minimal sedation level (RASS ≥ -1)
  * Have been monitored in intensive care for at least 24 hours
  * Have stable vital signs
  * Have no visual or auditory perception loss
  * Parental consent and verbal consent from the child must have been obtained

Exclusion Criteria:

* Severe neurological deficit or motor impairment

  * Severe pain, delirium, or agitation
  * Severe psychiatric diagnosis or requirement for high-dose sedation
  * Being in the terminal phase

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Level in Children | At baseline and immediately post-intervention
  State anxiety will be measured using the State Anxiety Inventory for Children, developed by Spielberger. The scale consists of 20 items assessing how children feel at the present moment, with total scores ranging from 20 to 80. Higher scores indicate higher levels of state anxiety. The Turkish version of the scale has demonstrated good reliability and validity in children and adolescents.
Respiratory Rate | At baseline and immediately post-intervention
  Respiratory rate will be measured as a physiological stress parameter using standard bedside monitoring systems routinely used in the pediatric intensive care unit. Respiratory rate will be recorded as breaths per minute.
Emotional Distress Level | At baseline and immediately post-intervention
  Emotional distress will be assessed using the Emotion Thermometer, a validated self-report tool adapted for use in Turkish children. Children will be asked to rate the intensity of five basic emotions (sadness, anxiety, fear, happiness, and calmness) on a numeric scale ranging from 0 (not experienced at all) to 10 (extremely intense). Higher scores indicate greater emotional intensity. The tool has demonstrated high internal consistency reliability.
Blood Pressure | At baseline and immediately post-intervention
  Systolic and diastolic blood pressure will be assessed non-invasively using standard bedside monitoring devices in the pediatric intensive care unit. Blood pressure values will be recorded in millimeters of mercury (mmHg).
Oxygen Saturation | At baseline and immediately post-intervention
  Oxygen saturation will be evaluated using pulse oximetry as part of routine bedside monitoring in the pediatric intensive care unit. Oxygen saturation values will be recorded as percentages (%)
Pain Intensity: | At baseline and immediately post-intervention
  Pain intensity be assessed using the Wong-Baker Faces Pain Rating Scale, a validated self-report measure appropriafor children based on age and communication ability. The scale allows children to indicate their level of pain using facial expressions.

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding the sharing of individual participant data has not yet been made. Any future data sharing will be considered following completion of the study, in accordance with ethical approval, participant consent, and applicable data protection regulations.

REFERENCES:
- [Background] 1. Amin, F. M., Ayed, M. M. A., & Mahmoud, N. F. (2022). Effect of Benson relaxation therapy on sleep quality among children in pediatric intensive care unit. International journal of health sciences, 6(S8), 6605-6619. 2. Apriany, D., Rakhmawati, W., Iskandarsyah, A., & Hilmanto, D. (2025). The Effect of The Mindfulness-Based Relaxation, Aromatherapy, and Prayer (RADO) Intervention on Anxiety and Quality of Life Among Children with Cancer. Journal of Multidisciplinary Healthcare, 1381-1392. 3. Bahcivan, O. & Eyrenci, A. (2018). The adaptation of Emotion Thermometer (ET) for Turkish speaking population. Psycho-Oncology 27: 215-216, 4. Bucur, S. M., Crișan, I. M., Cocoș, D. I., Bud, E. S., & Galea, C. (2025). Observational Study on Progressive Muscle Relaxation and Breathing Control for Reducing Dental Anxiety in Children. Medicina, 61(5), 876. 5. Ferro, M. M., Pegueroles, A. F., Lorenzo, R. F., Roy, M. Á. S., Forner, O. R., Jurado, C. M. E., ... & Alcaraz, A. B. (2023). The effect of a live music therapy intervention on critically ill paediatric patients in the intensive care unit: A quasi-experimental pretest-posttest study. Australian Critical Care, 36(6), 967-973. 6. Galinha, I. C., de Carvalho, J. L. D. C. S., de Oliveira, A. C. P., Arriaga, P., Gaspar, A. D., Silva, H. P., & Ortega, V. (2025). MindRegulation-SEL: randomized controlled trial of the effects of a relaxation and guided imagery intervention with socioemotional learning on the psychological and biophysiological well-being, socioemotional development, cognitive function and academic achievement of elementary school children. Trials, 26(1), 187. 7. Kalsotra, S., Froass, D., Gupta, A., Amaya, S., Tobias, J. D., & Olbrecht, V. A. (2025). Virtual Reality for Pediatric Postoperative Pain Management: Exploring Methods and Efficacy. Journal of Medical Internet Research, 27, e68348. 8. Köksal, Ö., Kilicarslan, E., & Emeksiz, S. (2025). Drawing and mutual storytelling to alleviate anxiety and improve emotional